CLINICAL TRIAL: NCT00568334
Title: Study of Two Formulations of GSK Biologicals' Varicella Vaccine Given as a 2-dose Course in the Second Year of Life
Brief Title: Study of Two Formulations of GSK Biologicals' Varicella Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109705
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-04

CONDITIONS: Varicella
Keywords: chickenpox; varicella; two-dose schedule; second year of life
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VARILRIX HSA-FREE GROUP (Experimental): Healthy male or female children between, and including, 11 and 21 months of age, who received 2 doses of Varilrix™ vaccine produced without human serum albumin (HSA-Free), administered subcutaneously into the deltoid region of the left upper arm, at Day 0 and Day 43-57 (Week 6).
  Interventions: Biological: Varilrix (inactivated varicella vaccine)
- VARILRIX GROUP (Experimental): Healthy male or female children between, and including, 11 and 21 months of age, who received 2 doses of Varilrix™ vaccine, administered subcutaneously into the deltoid region of the left upper arm, at Day 0 and Day 43-57 (Week 6).
  Interventions: Biological: Varilrix (inactivated varicella vaccine)

INTERVENTIONS:
Biological: Varilrix (inactivated varicella vaccine) — subcutaneously injection

SUMMARY:
The aim of this study is to evaluate a modified formulation of GSK Biologicals' live attenuated varicella vaccine. In vivo pre-clinical data show this change has no negative impact on vaccine safety. This present study is undertaken to rule out any negative impact on the immunogenicity and safety of GSK Biologicals' live attenuated varicella virus vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A male or female between, and including, 11 and 21 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days prior to the first study vaccine dose until 42 days after second study vaccine dose with the exception of oral polio vaccine (OPV) which can be given at any time and routine inactivated vaccines which can be administered up to eight days before each study vaccine dose.
* Previous vaccination against varicella.
* Known history of clinical varicella.
* Known exposure to varicella within 30 days prior to study start.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s), including systemic hypersensitivity to neomycin.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment. All vaccines can be administered to persons with a minor illness.
* Axillary temperature ≥ 37.5°C / Rectal temperature ≥ 38°C.
* Residence in the same household as a high risk person e.g.: new-born infants (0-4 weeks of age), pregnant women who have a negative history of chickenpox, persons with known immunodeficiency

Ages: 11 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2007-11-01 (Actual); Primary Completion 2008-03-18 (Actual); Study Completion 2008-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Czechia (2):
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Pardubice
- Hungary (6):
  - GSK Investigational Site, Bordány
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Zsombó

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Prymula R, Simko R, Povey M, Kulcsar A. Varicella vaccine without human serum albumin versus licensed varicella vaccine in children during the second year of life: a randomized, double-blind, non-inferiority trial. BMC Pediatr. 2016 Jan 13;16:7. doi: 10.1186/s12887-016-0546-5. PMID 26762528
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 109705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109705 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Started | 122 | 122
Completed | 121 | 121
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varilrix HSA-Free Group | Varilrix Group | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Continuous [Mean (Standard Deviation); unit: Months] | 15.6 (3.34) | 14.8 (3.08) | 15.20 (3.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 119
  Male | 63 | 62 | 125
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 122 | 122 | 244

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titers Against Varicella Zoster Virus (VZV)
Description: Antibody titers have been assessed by immunofluorescence assay (IFA) and presented as geometric mean titers (GMTs), for initially seronegative subjects [with anti-VZV titer below (<) 1:4].
Time Frame: At 43-57 days after the first vaccine dose (Week 6)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all eligible subjects who were seronegative for varicella antibodies at baseline and for whom pre-vaccination and post-vaccination serology results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 116 | 115
Titers | 172.6 [141.6 to 210.3] | 154.3 [128.7 to 185]
Statistical Analysis 1: Comparison: Varilrix HSA-Free Group vs Varilrix Group; Non-inferiority of Varilrix™ HSA-Free vaccine as compared to Varilrix™ vaccine in terms of geometric mean titers (GMTs) of varicella zoster virus (VZV) antibodies 43-57 days after the first vaccine dose; Test type: Non-Inferiority — The lower limit (LL) of the 95% confidence interval (CI) for the GMT ratio (derived from IFA) between Group Varilrix HSA-Free and (divided by) Group Varilrix is equal to or above (≥) the pre-defined clinical limit of 0.5; ANOVA; GMT Ratio = 1.12, 95% CI 2-sided [0.86 to 1.46]

2. Primary Outcome: Antibody Concentrations Against Varicella Zoster Virus (VZV)
Description: Antibody concentrations have been assessed by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL), for initially seronegative subjects [with anti-VZV concentration below (<) 25 mIU/mL].
Time Frame: At 43-57 days after the first vaccine dose (Week 6)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 116 | 115
mIU/mL | 123.5 [107.9 to 141.4] | 110.7 [98.4 to 124.6]
Statistical Analysis 1: Comparison: Varilrix HSA-Free Group vs Varilrix Group; Non-inferiority of Varilrix™ HSA-Free vaccine as compared to Varilrix™ vaccine in terms of geometric mean concentrations (GMCs) of varicella zoster virus (VZV) antibodies 43-57 days after the first vaccine dose; Test type: Non-Inferiority — The lower limit (LL) of the 95% confidence interval (CI) for the GMC ratio (derived from ELISA) between Group Varilrix HSA-Free and (divided by) Group Varilrix is equal to or above (≥) the pre-defined clinical limit of 0.67; ANOVA; GMC Ratio = 1.12, 95% CI 2-sided [0.93 to 1.33]

3. Secondary Outcome: Number of Seroconverted Subjects for Varicella Antibodies
Description: Seroconversion/seroresponse (considering the IFA data) was defined as the appearance of anti-VZV antibodies [i.e. titer/concentration greater than or equal to (≥) the assay cut-off value of 1:4] in the sera of subjects who were seronegative before vaccination.
Time Frame: At 43-57 days post-Dose 1 (Week 6) and 86-114 days post-Dose 2 (Week 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 116 | 115
Participants
  Anti-VZV, Week 6 | 114 | 114
  Anti-VZV, Week 12: number analyzed (Participants) | 115 | 112
  Anti-VZV, Week 12 | 115 | 112

4. Secondary Outcome: Number of Subjects With Anti-VZV Antibody Concentrations Above Cut-off Values
Description: Anti-VZV antibody concentrations greater than or equal to (≥) the assay cut-off values of: 25 mIU/mL, 50 mIU/mL and 75 mIU/mL have been assesssed by ELISA, in the sera of subjects who were seronegative before vaccination.
Time Frame: At 43-57 days post-Dose 1 (Week 6) and 86-114 days post-Dose 2 (Week 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 116 | 115
Participants
  Anti-VZV ≥ 25 mIU/mL, Week 6 | 114 | 113
  Anti-VZV ≥ 25 mIU/mL, Week 12: number analyzed (Participants) | 116 | 114
  Anti-VZV ≥ 25 mIU/mL, Week 12 | 116 | 114
  Anti-VZV ≥ 50 mIU/mL, Week 6 | 105 | 103
  Anti-VZV ≥ 50 mIU/mL, Week 12: number analyzed (Participants) | 116 | 114
  Anti-VZV ≥ 50 mIU/mL, Week 12 | 116 | 114
  Anti-VZV ≥ 75 mIU/mL, Week 6 | 89 | 89
  Anti-VZV ≥ 75 mIU/mL, Week 12: number analyzed (Participants) | 116 | 114
  Anti-VZV ≥ 75 mIU/mL, Week 12 | 116 | 114

5. Secondary Outcome: Antibody Titers Against Varicella Zoster Virus (VZV)
Description: as for outcome 1
Time Frame: At 86-114 days after the second vaccine dose (Week 12)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 115 | 112
Titers | 1452.5 [1240.7 to 1700.5] | 1395.4 [1183 to 1645.9]

6. Secondary Outcome: Antibody Concentrations Against Varicella Zoster Virus (VZV)
Description: as for outcome 2
Time Frame: At 86-114 days after the second vaccine dose (Week 12)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 116 | 114
mIU/mL | 1013.6 [880.9 to 1166.4] | 999.2 [877.3 to 1138.1]

7. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = incidence of a particular symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 121 | 122
Participants
  Any Pain, Dose 1 | 13 | 15
  Grade 3 Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 33 | 34
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 5 | 7
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 121 | 121
  Any Pain, Dose 2 | 23 | 18
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 121 | 121
  Grade 3 Pain, Dose 2 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 121 | 121
  Any Redness, Dose 2 | 44 | 46
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 121 | 121
  Grade 3 Redness, Dose 2 | 6 | 3
  Any Swelling, Dose 2: number analyzed (Participants) | 121 | 121
  Any Swelling, Dose 2 | 18 | 14
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 121 | 121
  Grade 3 Swelling, Dose 2 | 2 | 2

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fever [defined as axillary fever ≥ 37.5 degrees Celsius (°C)] and generalized rash. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 fever = temperature above (>) 39.0°C after vaccination. Grade 3 rash = more than (>) 150 lesions. Related = considered by the investigator to be causally related to the study vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period following each dose
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 121 | 122
Participants
  Any Temperature, Dose 1 | 64 | 52
  Grade 3 Temperature, Dose 1 | 13 | 11
  Related Temperature, Dose 1 | 2 | 2
  Any Rash, Dose 1 | 1 | 0
  Grade 3 Rash, Dose 1 | 54 | 53
  Related Rash, Dose 1 | 6 | 12
  Any Temperature, Dose 2: number analyzed (Participants) | 121 | 121
  Any Temperature, Dose 2 | 3 | 3
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 121 | 121
  Grade 3 Temperature, Dose 2 | 1 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 121 | 121
  Related Temperature, Dose 2 | 31 | 18
  Any Rash, Dose 2: number analyzed (Participants) | 121 | 121
  Any Rash, Dose 2 | 0 | 0
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 121 | 121
  Grade 3 Rash, Dose 2 | 31 | 23
  Related Rash, Dose 2: number analyzed (Participants) | 121 | 121
  Related Rash, Dose 2 | 1 | 0

9. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Event (AE)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within the 43-day (Days 0-42) post-vaccination period following each dose
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 122 | 122
Participants
  Any AE(s), Dose 1 | 56 | 45
  Any AE(s), Dose 2: number analyzed (Participants) | 121 | 121
  Any AE(s), Dose 2 | 35 | 42

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that results in death, are life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to study end (Day 86-114)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
Number analyzed (Participants) | 122 | 122
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: Solicited local symptoms: during the 4-day (Days 0-3) post each dose. Solicited general symptoms and unsolicited AEs: during the 43-day (Days 0-42) post each dose. SAEs: during the entire study period (Day 0 to Day 86/114).
Arm/Group | Varilrix HSA-Free Group | Varilrix Group
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/122
Serious Adverse Events (participants affected / at risk) | 2/122 | 5/122
Other Adverse Events (participants affected / at risk) | 103/122 | 100/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varilrix HSA-Free Group (N=122) | Varilrix Group (N=122)
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Breath holding (Psychiatric disorders) | 0 | 1
Otitis media (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Varilrix HSA-Free Group (N=122) | Varilrix Group (N=122)
Pain (Dose 1) (General disorders) | 13/121 | 15
Redness (Dose 1) (General disorders) | 33/121 | 34
Swelling (Dose 1) (General disorders) | 5/121 | 7
Pain (Dose 2) (General disorders) | 23/121 | 18/121
Redness (Dose 2) (General disorders) | 44/121 | 46/121
Swelling (Dose 2) (General disorders) | 18/121 | 14/121
Fever (Dose 1) (General disorders) | 64/121 | 52
Fever (Dose 2) (General disorders) | 54/121 | 53/121
Bronchitis (Dose 1) (Infections and infestations) | 15 | 8
Viral infection (Dose 1) (Infections and infestations) | 11 | 11
Rhinitis (Dose 1) (Infections and infestations) | 6 | 8
Bronchitis (Dose 2) (Infections and infestations) | 8/121 | 11/121
Viral infection (Dose 2) (Infections and infestations) | 6/121 | 13/121
Rhinitis (Dose 2) (Infections and infestations) | 7/121 | 1/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.